CLINICAL TRIAL: NCT05242666
Title: Evaluating Advanced Imaging Techniques for Use in the Assessment of Degenerative Cervical Myelopathy
Brief Title: Quantiative MRI and Myelin-PET for the Assessment of Degenerative Cervical Myelopathy
Acronym: IMAGE-DCM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Wolfson Brain Imaging Centre (Unknown)
Responsible Party: Principal Investigator, Benjamin Davies, Honorary Specialist Registrar, Department of Neurosurgery, Cambridge University Hospital, Cambridge University Hospitals NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 274826
Record Dates: First submitted 2019-12-05; First posted 2022-02-16 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Cervical Spondylosis With Myelopathy; Degenerative Cervical Myelopathy
Keywords: Positron Emission Tomography; Magnetic Resonance Imaging
MeSH Terms: interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Intervention Model Description: Observational study of patients undergoing surgery for degenerative cervical myelopathy, allocated to receive an additional form of imaging assessment before and after surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DCM1: MRI Spinal Cord (Other): 3T MR Imaging of the cervical spinal cord, before and at 3-6 months after surgery.
  Interventions: Diagnostic Test: 3T MR Imaging of the cervical spinal cord
- DCM2: MRI Brain and Spinal Cord (Other): 3T MR Imaging of the brain and cervical spinal cord, before and at 3-6 months after surgery. A subset will also be invited to undergo 7T MRI Brain and Spinal Cord Imaging.
  Interventions: Diagnostic Test: 3T MR Imaging of the cervical spinal cord; Other: 3T MR Imaging of the Brain; Other: 7T MR Imaging of the Spinal Cord
- DCM3: [11C]-PIB MR/PET Cervical Spinal Cord (Other): [11C]PIB PET/MR Imaging of the cervical spinal cord, before and at 3-6 months after surgery.
  Interventions: Other: Positron Emission Tomography using [11C]PIB
- Healthy Volunteer: MRI Brain and Spinal Cord (Other): Age-Matched Healthy Controls will undergo MRI Brain and Spinal Cord. A subset will also be invited to undergo interval imaging at 3-6 months.
  Interventions: Diagnostic Test: 3T MR Imaging of the cervical spinal cord; Other: 3T MR Imaging of the Brain

INTERVENTIONS:
Diagnostic Test: 3T MR Imaging of the cervical spinal cord — Patients will undergo either Magnetic Resonance Imaging of the Spinal Cord
  Arms: DCM1: MRI Spinal Cord; DCM2: MRI Brain and Spinal Cord; Healthy Volunteer: MRI Brain and Spinal Cord
Other: Positron Emission Tomography using [11C]PIB — Patients will undergo combination MRI/PET using a [11C]PIB radiotracer
  Arms: DCM3: [11C]-PIB MR/PET Cervical Spinal Cord
Other: 3T MR Imaging of the Brain — 3T MR Imaging of the Brain
  Arms: DCM2: MRI Brain and Spinal Cord; Healthy Volunteer: MRI Brain and Spinal Cord
Other: 7T MR Imaging of the Spinal Cord — 7T MR Imaging of the Spinal Cord
  Arms: DCM2: MRI Brain and Spinal Cord

SUMMARY:
To use advanced imaging techniques, including MRI Brain and Spinal Cord, and MRI/PET Spinal Cord to provide an assessment of Degenerative Cervical Myelopathy to improve understanding of the pathophysiology and natural history of DCM.

DETAILED DESCRIPTION:
Degenerative Cervical Myelopathy (DCM) is a disabling condition affecting up to 2% of adults. It arises when arthritic changes in the cervical spine compress and injure the spinal cord, causing progressive loss of bodily function.

Surgery will remove compression and stop injury. However, for a full recovery, it must occur before irreversible spinal cord damage. Current assessments cannot provide this information and today, 95% of patients are left disabled: an assessment that measures spinal cord damage would change this tomorrow.

Imaging advances, well established for measuring disease of the brain, have the potential to provide this in DCM, but requires further investigation. This is the subject of this proposed application: specifically, to investigate 3 different but promising imaging approaches for the assessment of DCM:

1. Advanced magnetic resonance imaging (MRI) to image within the spinal cord
2. Advanced MRI to measure the changes that occur within the brain following DCM
3. Positron Emission Tomography (PET) to measure the active disease biology within the spinal cord.

Individuals with a diagnosis of DCM, will be invited to undergo one of these options, before and after their surgical treatment. Clinical measures used in routine practice will be noted, in order to draw comparisons with imaging. A healthy control group will also be used for MRI imaging, in order to identify changes specific to DCM. Aside from the additional imaging, there will be no changes in routine care.

ELIGIBILITY:
Inclusion Criteria

1. Participant has a diagnosis of DCM, based on a combination of symptoms, signs and conventional MRI findings (Table 2)
2. Participant is scheduled for surgical treatment for DCM
3. Participant is willing and able to give informed consent for participation in the study;
4. Male or Female, aged 18 - 85 years (inclusive);

Exclusion Criteria

The participant may not enter the study if ANY of the following apply:

1. Participant unable to give informed consent;
2. Participant unable to undergo, or intolerant of MR or PET/MR imaging
3. Participant has co-existing or prior neurological disease of the brain, spinal cord, or peripheral nervous system, including but not limited to, Lumbar Canal Stenosis, Multiple Sclerosis, Dementia and Parkinson's Disease.
4. Contraindications to MRI: These are chiefly the presence of metallic implants that are not known to be MR safe, particularly in terms of movement or substantial heating. Devices that may need to be considered in this context include (this is not an exhaustive list, and this issue will be considered on a case-by-case basis for any implant or external fixation device):

   * Cerebral aneurysm clips not known to be MR safe
   * Intra-ocular metallic shards
   * Cochlear implants
   * Automatic cardioverter defibrillators
   * Nerve stimulation units
   * Other electronic implants, such as cardiac pacemakers
   * Orthopedic external fixations

Exclusion Criteria Specific for PET/MR Imaging Stream

In addition, the following exclusion criteria will apply for PET imaging, to reduce implications of exposure to ionising radiation, or interpretation of findings.

1. Female patients who are pregnant or breast-feeding
2. Participants whose DCM surgery will include the insertion of metallic implants to secure multiple levels of the spine (technically termed 'instrumentation')
3. Age <40

4.3.2 Volunteers

Inclusion Criteria

1. Participant is willing and able to give informed consent for participation in the study;
2. Male or Female, aged 18 - 85 years (inclusive); Exclusion Criteria

The participant may not enter the study if ANY of the following apply:

1. Participant unable to give informed consent;
2. Participant unable to undergo, or intolerant of MR imaging
3. Participant has co-existing or prior neurological disease of the brain, spinal cord, or peripheral nervous system, including but not limited to, Lumbar Canal Stenosis, Multiple Sclerosis, Dementia and Parkinson's Disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-17 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Modified Japanese Orthopaedics Association (mJOA) | 6 Months Post Surgery

SECONDARY OUTCOMES:
Short-Form 36 (SF-36) | Routine Clinical Care: Baseline and 3-6 Months Post-Operatively
  Quality of Life (0-100, where 50 is normal for geographical population. Higher score is better)
Numeric Rating Scale (NRS) Pain | Routine Clinical Care: Baseline and 3-6 Months Post-Operatively
  Pain Score (0-10, where 10 is maximum pain, and 0 is no pain. Lower score is better)
Myelopathy.org Symptom Inventory [MOSI] | Routine Clinical Care: Baseline and 3-6 Months Post-Operatively
  Quality of Life and Disease Specific Measure (Range of Myelopathy symptoms are scored as Not present, on an intensity scale of 0 to 10, where 10 is worse).
Neurological Exam | Routine Clinical Care: Baseline and 3-6 Months Post-Operatively
  Routine Neurological Exam (Motor and Sensory changes to hands, arms and legs, long-tract signs in cluded reflexes, Hoffman's and Babbinski's reflexes)

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Annoymised Data will be made available, for collaboration, at the discretion of the senior investigators upon completion of the study.

REFERENCES:
- [Background] Davies BM, Mowforth OD, Smith EK, Kotter MR. Degenerative cervical myelopathy. BMJ. 2018 Feb 22;360:k186. doi: 10.1136/bmj.k186. No abstract available. PMID 29472200